CLINICAL TRIAL: NCT00460018
Title: Diet, Exercise and Breastfeeding Intervention (DEBI) Program for Women With Gestational Diabetes
Brief Title: Diet, Exercise, and Breastfeeding Intervention Program for Women With Gestational Diabetes (DEBI Trial)
Acronym: DEBI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Assiamira Ferrara, MD PhD, Kaiser Permanente Division of Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CN-04AFerr-04-H; CN-03AFerr-02
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2009-06-19 (Estimated); Status verified 2009-01

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Gestational Diabetes Mellitus; Weight Loss; Physical Activity; Breastfeeding; Pregnancy; Postpartum; Intervention; Prevention
MeSH Terms: conditions — Diabetes, Gestational; Weight Loss; Motor Activity; Breast Feeding | interventions — Diet; Exercise; Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Women receiving the DEBI Intervention
  Interventions: Behavioral: Diet, Exercise, and Breastfeeding Intervention
- No intervention (No Intervention): Women receiving standard care

INTERVENTIONS:
Behavioral: Diet, Exercise, and Breastfeeding Intervention — Phase I (Pregnancy Program from GDM diagnosis to delivery): One in-person session with the lifestyle coach, two phone calls with the lifestyle coach, and one in-person session with the lactation consultant
  Phase II (Early Post-partum Period from delivery to 6 weeks post-partum): Two to four routine phone calls with the lactation consultant
  Phase III (Late Post-partum Period 6 weeks to 7 months postpartum): Two in-person sessions with the lifestyle coach, up to 11 phone calls with the lifestyle coach, and two to three routine calls with the lactation consultant
  Phase IV (Maintenance Phase 8 months to 1 year postpartum): One newsletter from the lifestyle coaches, two recipe letters and continue calls with the lifestyle coach (optional)
  Other Names: Intervention
  Arms: Intervention

SUMMARY:
The primary aim of this study is to evaluate whether a lifestyle intervention of diet, exercise, and breastfeeding is associated with decreased postpartum weight retention and reduced plasma glucose levels, measured at 6-weeks and 1-year postpartum, among women with gestational diabetes mellitus (GDM). Secondary outcomes are postpartum levels of plasma insulin, markers of insulin resistance, adiponectin, dietary fat, physical activity, and breastfeeding duration.

DETAILED DESCRIPTION:
Postpartum predictors of type 2 diabetes incidence in women with GDM are pregnancy weight retention and postpartum weight gain. By promoting physical activity and appropriate diet during pregnancy and soon after delivery, and preventing excessive pregnancy weight gain and postpartum weight retention, the postpartum incidence of obesity and type 2 diabetes might be reduced or delayed in GDM women. We are implementing and evaluating a lifestyle intervention of diet, physical activity, and breastfeeding among women with GDM. The diet and physical activity elements of the intervention are similar to the DPP-Follow-up study. All participants have GDM by plasma glucose levels measured during a standard 100-g, 3-h OGTT according to the ADA and the ACOG criteria and have no contraindications to participating in a diet and physical activity program. At study entry, eligible women are randomly assigned to life-style intervention or usual medical care. The intervention starts during pregnancy and continues for one year postpartum. It consists of structured, individually tailored, in-person sessions and telephone calls with a lactation consultant and a life-style coach. The goals of the intervention during pregnancy are to help GDM women comply with the Institute of Medicine guidelines for weight gain by following the ADA and ACOG recommendations for physical activity and diet. After pregnancy, the goals of the intervention are to help women exclusively breastfeed for at least six months and reach their pre-pregnancy weight. For those women who were overweight or obese prior to pregnancy, the additional goal of a reduction in weight of at least 5% of their pre-pregnancy weight is also set. For the maintenance phase of the intervention, beginning at 8 months postpartum, the intervention women receive tailored written materials in the mail and telephone calls reinforcing the positive changes they have adopted. All participants have follow-up clinic visits at 8-week, 8-month, 12-month, 18-month, and 24-month after delivery. Data analyses will be by intent-to-treat. Demographics, psychosocial and behavioral factors that may be related to success at achieving the postpartum weight goals and the secondary postpartum outcomes will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Gestational Diabetes Mellitus

Exclusion Criteria:

* Ever diagnosed with diabetes when not pregnant
* Ever diagnosed with cardiovascular disease
* Ever diagnosed with lung disease
* Hemoglobin < 9.5 mg/dl
* Hematocrit less than 30%
* SBP >= 140 or DBP >= 90 in the last month
* Diagnosis of thyroid disease in the last month

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2005-09

PRIMARY OUTCOMES:
Postpartum weight retention | no more than 1.5 years

SECONDARY OUTCOMES:
reduced plasma glucose levels (measured at 6 weeks and 1 year postpartum) | 1 year
levels of plasma insulin | 1 year
markers of insulin resistance | 1 year
adiponectin | 1 year
dietary fat | no more than 1.5 years
physical activity | no more than 1.5 years
breastfeeding duration | no more than 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Assiamira Ferrara, MD, PhD, Principal Investigator — Kaiser Permanente Division of Research
Locations (5):
- United States (5):
  - Kaiser Permanente Oakland, Oakland, California
  - Kaiser Permanente Division of Research, Oakland, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - Kaiser Permanente Santa Clara/Santa Teresa, Santa Clara, California
  - Kaiser Permanente Walnut Creek, Walnut Creek, California

REFERENCES:
- [Background] Metzger BE. Summary and recommendations of the Third International Workshop-Conference on Gestational Diabetes Mellitus. Diabetes. 1991 Dec;40 Suppl 2:197-201. doi: 10.2337/diab.40.2.s197. No abstract available. PMID 1748259
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] O'Toole ML, Sawicki MA, Artal R. Structured diet and physical activity prevent postpartum weight retention. J Womens Health (Larchmt). 2003 Dec;12(10):991-8. doi: 10.1089/154099903322643910. PMID 14709187
- [Background] Leermakers EA, Anglin K, Wing RR. Reducing postpartum weight retention through a correspondence intervention. Int J Obes Relat Metab Disord. 1998 Nov;22(11):1103-9. doi: 10.1038/sj.ijo.0800734. PMID 9822949
- [Derived] Ferrara A, Hedderson MM, Albright CL, Ehrlich SF, Quesenberry CP Jr, Peng T, Feng J, Ching J, Crites Y. A pregnancy and postpartum lifestyle intervention in women with gestational diabetes mellitus reduces diabetes risk factors: a feasibility randomized control trial. Diabetes Care. 2011 Jul;34(7):1519-25. doi: 10.2337/dc10-2221. Epub 2011 May 3. PMID 21540430